CLINICAL TRIAL: NCT02259088
Title: A 12-month, Randomized, Double-masked, Multicenter, Laser-controlled Phase III Study Assessing the Efficacy and Safety of 0.5 mg Ranibizumab Dosed PRN in Subjects With Visual Impairment Due to Diabetic Macular Edema in Chinese Patients
Brief Title: A 12-month, Randomized, Efficacy and Safety Study of 0.5 mg Ranibizumab vs Laser in Chinese Diabetic Macular Edema (DME) Patients
Acronym: REFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRFB002D2305
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Macular Edema; Visual Impairment
Keywords: DME; macular edema; vision impairment; Chinese; diabetes
MeSH Terms: conditions — Vision Disorders; Macular Edema; Diabetes Mellitus | interventions — Ranibizumab; Lasers; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab (RFB002) (Experimental): 3 initial intravitreal injections to the study eye at Day 1, Month 1 and Month 2, followed by as-needed intravitreal injections of ranibizumab 0.5 mg guided by VA stabilization, plus sham laser
  Interventions: Drug: Ranibizumab (RFB002); Procedure: Sham laser
- Laser (Active Comparator): Laser photocoagulation applied to the study eye at Day 1, followed by active laser photocoagulation at intervals no shorter than 3 months apart, plus sham injections
  Interventions: Procedure: Laser; Drug: Sham injection

INTERVENTIONS:
Drug: Ranibizumab (RFB002) — Ranibizumab 0.5 mg/0.05 mL for intravitreal injection
  Other Names: Lucentis
  Arms: Ranibizumab (RFB002)
Procedure: Laser — Laser photocoagulation according to Early Treatment Diabetic Retinopathy Study (ETDRS) guidelines
  Arms: Laser
Drug: Sham injection — Imitation of an intravitreal injection consisting of an empty vial and an injection syringe without a needle
  Arms: Laser
Procedure: Sham laser — Imitation of an active laser
  Arms: Ranibizumab (RFB002)

SUMMARY:
Study of efficacy and safety of 0.5 mg ranibizumab in Chinese patients with diabetic macular edema (DME)

DETAILED DESCRIPTION:
The purpose of this study was to provide efficacy and safety data on 0.5 mg ranibizumab intravitreal injections compared to laser photocoagulation in Chinese patients with visual impairment due to DME. Treatment was driven by achieving vision stabilization.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female Chinese patients ≥ 18 years of age with diabetes mellitus and with HbA1c ≤10.0%
* Stable medication for diabetes within 3 months prior to Visit 1
* Visual impairment due to DME with BCVA score between 78 and 39 letters as measured by ETDRS-like charts at 4 meters

Key Exclusion Criteria:

* Stroke or myocardial infarction less than 3 months prior to screening visit
* Uncontrolled hypertension
* Active ocular infection or intraocular inflammation in any eye
* Treatment with any anti-angiogenic drugs within 3 months prior to baseline visit in any eye
* Active proliferative diabetic retinopathy in study eye
* Use of other investigational drugs within 30 days and systemic anti-VEGF drugs within 6 months prior to baseline visit
* Prior laser photocoagulation or intraocular procedure within 3 months prior to baseline in study eye
* History of intravitreal corticosteroid treatment in phakic study eye, and in aphakic or pseudophakic within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- China (17):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After eligibility confirmation, patients were randomized in a 4:1 ratio to 2 treatment arms.
Period: Overall Study
Arm/Group | Ranibizumab (RFB002) | Laser
Started (All randomized participants) | 307 | 77
Full Analysis Set | 307 | 77
Treated (Safety Analysis Set) | 307 | 75
Completed | 279 | 63
Not Completed | 28 | 14
Not completed — Adverse Event | 6 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 2 | 0
Not completed — Physician Decision | 5 | 2
Not completed — Protocol deviation | 5 | 0
Not completed — Subject/guardian decision | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab (RFB002) | Laser | Total
Number analyzed (Participants) | 307 | 77 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (8.70) | 59.0 (9.19) | 58.7 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 38 | 206
  Male | 139 | 39 | 178
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: letters] — Visual acuity with eyeglasses was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at an initial testing distance of 4 meters. A letter score was calculated based on the number of letters correctly identified at the specified distance. One eye (study eye) contributed to the analysis.
  letters | 59.6 (10.53) | 58.2 (9.43) | 59.3 (10.32)

OUTCOME MEASURES:

1. Primary Outcome: Mean Average Change From Baseline in Best-Corrected Visual Acuity (BCVA) (Letters) to Month 1 Through 12
Description: Visual acuity with eyeglasses was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at an initial testing distance of 4 meters. A letter score was calculated based on the number of letters correctly identified at the specified distance. Twelve monthly BCVA values were averaged [(Month1+Month2+...+Month12)/12], and the baseline BCVA value was subtracted from the average. A positive change value indicates an improvement in visual acuity, while a negative change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Monthly from Month 1 through Month 12
Population: Full Analysis Set (FAS). Missing values imputed by the mean value last observation carried forward (MV-LOCF).
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 303 | 75
letters | 6.8 (6.58) | 1.1 (7.73)
Statistical Analysis 1: Comparison: Ranibizumab (RFB002) vs Laser; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; One-sided p-value for treatment difference is derived from the two-sided stratified Cochran-Mantel-Haenszel test using the row means score statistics; Least Squares Mean Difference = 5.8, 95% CI 2-sided [4.1 to 7.5] — Estimated from ANOVA (stratified) model. Stratified analysis includes DME type (focal, diffuse, honeycomb and petaloid) and Baseline BCVA(≤ 60 letters and > 60 letters) as factors

2. Secondary Outcome: Mean Change From Baseline in BCVA (Letters) at Each Visit
Description: Visual acuity with eyeglasses was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at an initial testing distance of 4 meters. A letter score was calculated based on the number of letters correctly identified at the specified distance. A positive change value indicates an improvement in visual acuity, while a negative change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Monthly from Month 1 through Month 12
Population: Full Analysis Set (FAS) with missing values imputed by the last observation carried forward (LOCF). The number analyzed is the number of patients with a value for both baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 303 | 75
letters
  Change from Baseline at Month 1: number analyzed (Participants) | 301 | 75
  Change from Baseline at Month 1 | 4.0 (5.59) | -0.9 (5.50)
  Change from Baseline at Month 2 | 5.8 (6.44) | 0.0 (8.08)
  Change from Baseline at Month 3 | 6.9 (6.91) | 1.1 (9.18)
  Change from Baseline at Month 4 | 6.6 (7.23) | 0.0 (11.64)
  Change from Baseline at Month 5 | 6.8 (7.41) | 0.6 (10.61)
  Change from Baseline at Month 6 | 6.8 (8.00) | 0.3 (11.01)
  Change from Baseline at Month 7 | 6.8 (7.95) | 1.3 (10.13)
  Change from Baseline at Month 8 | 7.4 (8.12) | 1.9 (9.69)
  Change from Baseline at Month 9 | 7.3 (8.18) | 1.8 (9.33)
  Change from Baseline at Month 10 | 7.2 (8.45) | 1.6 (9.23)
  Change from Baseline at Month 11 | 7.8 (8.55) | 1.7 (9.35)
  Change from Baseline at Month 12 | 7.8 (8.72) | 2.5 (8.78)

3. Secondary Outcome: Mean Change From Baseline in Central Sub-Field Thickness (CSFT) at Each Visit
Description: CSFT (the average retinal thickness of the circular area within 1 millimeter diameter around the foveal center) was assessed using Optical Coherence Tomography (OCT). A negative change value indicates an improvement in macular edema, while a positive change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Monthly from Month 1 through Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 301 | 75
micrometers
  Change from Baseline at Month 1: number analyzed (Participants) | 299 | 75
  Change from Baseline at Month 1 | -126.7 (140.59) | -33.1 (113.34)
  Change from Baseline at Month 2 | -141.3 (146.15) | -48.8 (133.22)
  Change from Baseline at Month 3 | -154.2 (147.94) | -58.5 (157.30)
  Change from Baseline at Month 4 | -130.4 (152.60) | -72.6 (149.13)
  Change from Baseline at Month 5 | -141.0 (153.28) | -72.3 (150.45)
  Change from Baseline at Month 6 | -146.2 (154.87) | -72.9 (152.47)
  Change from Baseline at Month 7 | -138.4 (161.04) | -72.4 (150.86)
  Change from Baseline at Month 8 | -146.9 (154.68) | -81.8 (151.89)
  Change from Baseline at Month 9 | -142.4 (156.03) | -80.9 (157.69)
  Change from Baseline at Month 10 | -137.6 (152.73) | -82.9 (166.16)
  Change from Baseline at Month 11 | -144.8 (159.87) | -88.1 (170.11)
  Change from Baseline at Month 12 | -146.5 (157.61) | -85.9 (166.60)

4. Secondary Outcome: Percentage of Patients With BCVA Gain of ≥ 10 and ≥ 15 Letters From Baseline at Month 12
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS) with missing values imputed by the last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 303 | 75
percentage of participants
  Gain of ≥ 10 letters | 40.6 | 20.0
  Gain of ≥ 15 letters | 18.5 | 8.0

5. Secondary Outcome: Percentage of Patients With BCVA Loss of < 10 and < 15 Letters From Baseline to Month 12
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS) with missing values imputed by the last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 303 | 75
percentage of participants
  Loss of < 10 letters | 97.0 | 89.3
  Loss of <15 letters | 99.0 | 97.3

6. Secondary Outcome: Percentage of Patients With BCVA ≥ 73 Letters at Month 12
Description: Visual acuity with eyeglasses was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at an initial testing distance of 4 meters. A letter score was calculated based on the number of letters correctly identified at the specified distance. A positive change value indicates an improvement in visual acuity, while a negative change value indicates a worsening. BCVA ≥ 73 letters is approximately equivalent to 20/40 on a Snellen chart. One eye (study eye) contributed to the analysis.
Time Frame: Month 12
Population: Full Analysis Set (FAS) with missing values imputed by the last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 303 | 75
percentage of participants | 36.0 | 21.3

7. Secondary Outcome: Mean Average Change in BCVA From Month 4 to Month 12 Compared to Month 3
Description: Visual acuity with eyeglasses was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at an initial testing distance of 4 meters. A letter score was calculated based on the number of letters correctly identified at the specified distance. Nine monthly BCVA values were averaged [(Month4+Month5+...+Month12)/9],and the Month 3 BCVA value was subtracted from the average. A positive change value indicates an improvement in visual acuity, while a negative change value indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Monthly from Month 3 through Month 12
Population: Full Analysis Set (FAS) with missing values imputed by the last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 303 | 75
letters
  Month 3 | 66.4 (10.66) | 59.2 (12.63)
  Average Change from Baseline Month 4 to Month 12 | 0.3 (4.51) | 0.2 (6.08)

8. Secondary Outcome: Mean Change From Baseline in Patient-Reported Visual Functioning at Month 6 and Month 12, Composite Score
Description: Visual functioning was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in visual functioning, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: Full Analysis Set, observed data (no missing data imputations). The number analyzed is the number of patients with a value for both baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | 2.5 (13.54) | 0.5 (13.17)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | 0.6 (14.99) | -0.4 (15.89)

9. Secondary Outcome: Mean Change From Baseline in Patient-Reported General Health at Month 6 and Month 12
Description: General health was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in general health, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | -1.5 (22.32) | -0.4 (21.81)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | -2.3 (24.34) | -4.3 (26.56)

10. Secondary Outcome: Mean Change From Baseline in Patient-Reported General Vision at Month 6 and Month 12
Description: General vision was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in general vision, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | 6.2 (18.77) | 4.7 (19.58)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | 5.9 (18.12) | 5.9 (20.06)

11. Secondary Outcome: Mean Change From Baseline in Patient-Reported Color Vision at Month 6 and Month 12
Description: Color vision was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in color vision, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: Full Analysis Set, observed data (no missing data imputations).The number analyzed is the number of patients with a value for both baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 280 | 67
units on a scale
  Change from Baseline at Month 6 | 2.0 (16.68) | 2.2 (17.26)
  Change from Baseline at Month 12: number analyzed (Participants) | 262 | 61
  Change from Baseline at Month 12 | 0.2 (21.55) | 1.6 (20.35)

12. Secondary Outcome: Mean Change From Baseline in Patient-Reported Peripheral Vision at Month 6 and Month 12
Description: Peripheral vision was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in peripheral vision, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 291 | 68
units on a scale
  Change from Baseline at Month 6 | 1.4 (20.51) | 5.5 (22.38)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | -2.3 (25.07) | 3.1 (27.64)

13. Secondary Outcome: Mean Change From Baseline in Patient-Reported Ocular Pain at Month 6 and Month 12
Description: Ocular pain was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in ocular pain, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | -1.5 (20.71) | 1.5 (20.89)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | -0.3 (19.89) | 4.1 (22.72)

14. Secondary Outcome: Mean Change From Baseline in Patient-Reported Near Activities at Month 6 and Month 12
Description: Near activities were assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in near activities, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 291 | 68
units on a scale
  Change from Baseline at Month 6 | 5.6 (23.81) | -1.7 (24.20)
  Change from Baseline at Month 12: number analyzed (Participants) | 278 | 64
  Change from Baseline at Month 12 | 0.6 (24.64) | -3.4 (21.93)

15. Secondary Outcome: Mean Change From Baseline in Patient-Reported Distance Activities at Month 6 and Month 12
Description: Distance activities were assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in distance activities, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | 5.4 (20.79) | -2.8 (19.35)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | 1.6 (23.74) | -5.5 (21.89)

16. Secondary Outcome: Mean Change From Baseline in Patient-Reported Social Functioning at Month 6 and Month 12
Description: Social functioning was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in social functioning, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 67
units on a scale
  Change from Baseline at Month 6 | 2.1 (19.24) | -1.5 (15.31)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 63
  Change from Baseline at Month 12 | -0.8 (21.58) | -3.2 (18.51)

17. Secondary Outcome: Mean Change From Baseline in Patient-Reported Mental Health at Month 6 and Month 12
Description: Mental health was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in mental health, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | 1.8 (23.07) | -0.2 (23.58)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | 1.3 (25.05) | 0.6 (23.32)

18. Secondary Outcome: Mean Change From Baseline in Patient-Reported Roles Difficulties at Month 6 and Month 12
Description: Roles difficulties were assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in roles difficulties, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | 1.4 (27.05) | -0.4 (24.24)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | 0.4 (27.62) | -1.4 (28.36)

19. Secondary Outcome: Mean Change From Baseline in Patient-Reported Dependency at Month 6 and Month 12
Description: Dependency was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in dependency, while a negative change value indicates a worsening.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 292 | 68
units on a scale
  Change from Baseline at Month 6 | 0.2 (27.95) | -4.3 (27.53)
  Change from Baseline at Month 12: number analyzed (Participants) | 279 | 64
  Change from Baseline at Month 12 | 0.9 (30.47) | -5.3 (27.87)

20. Secondary Outcome: Mean Change From Baseline in Patient-Reported Driving at Month 6 and Month 12
Description: Driving was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in driving, while a negative change value indicates a worsening. Note: Many patients did not answer the driving related question as they did not drive at all.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab (RFB002) | Laser
Number analyzed (Participants) | 44 | 12
units on a scale
  Change from Baseline at Month 6 | 2.8 (15.87) | 2.8 (20.52)
  Change from Baseline at Month 12: number analyzed (Participants) | 41 | 11
  Change from Baseline at Month 12 | -0.2 (12.29) | 4.5 (27.98)

21. Secondary Outcome: Mean Number of Ranibizumab Re-treatments Received in the Study Eye From Month 3 Onward
Description: A ranibizumab re-treatment was defined as an administration of ranibizumab injection at a scheduled visit following at least one non-missed visit where ranibizumab was not administered in the study eye due to visual acuity stabilization. This outcome measure was pre-specified for the Ranibizumab 0.5 mg arm only.
Time Frame: Monthly from Month 3 through Month 12
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: retreatments
Arm/Group | Ranibizumab (RFB002)
Number analyzed (Participants) | 301
retreatments | 1.6 (0.64)

ADVERSE EVENTS:
Time Frame: Day 1 through study completion, an average of 1 year
Arm/Group | Ranibizumab (RFB002) | Laser
Serious Adverse Events (participants affected / at risk) | 57/307 | 15/75
Other Adverse Events (participants affected / at risk) | 116/307 | 30/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (RFB002) (N=307) | Laser (N=75)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Cataract (Fellow eye) (Eye disorders) | 2 | 0
Cataract (Study eye) (Eye disorders) | 1 | 0
Diabetic retinal oedema (Fellow eye) (Eye disorders) | 1 | 2
Diabetic retinopathy (Fellow eye) (Eye disorders) | 1 | 0
Eye haemorrhage (Fellow eye) (Eye disorders) | 1 | 0
Glaucoma (Fellow eye) (Eye disorders) | 1 | 0
Retinal detachment (Fellow eye) (Eye disorders) | 0 | 1
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 3 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Conjunctivitis viral (Fellow eye) (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal flattening (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basilar artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 4 | 0
Diabetic neuropathy (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 5 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal arteriosclerosis (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic dermopathy (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2
Diabetic vascular disorder (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (RFB002) (N=307) | Laser (N=75)
Anaemia (Blood and lymphatic system disorders) | 10 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 11 | 1
Dry eye (Fellow eye) (Eye disorders) | 10 | 1
Dry eye (Study eye) (Eye disorders) | 11 | 1
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 11 | 3
Vitreous haemorrhage (Study eye) (Eye disorders) | 5 | 3
Nasopharyngitis (Infections and infestations) | 20 | 7
Upper respiratory tract infection (Infections and infestations) | 26 | 2
Urinary tract infection (Infections and infestations) | 15 | 3
Alanine aminotransferase increased (Investigations) | 3 | 4
Intraocular pressure increased (Study eye) (Investigations) | 16 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 | 3
Diabetic nephropathy (Renal and urinary disorders) | 10 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 2
Hypertension (Vascular disorders) | 17 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.